CLINICAL TRIAL: NCT01435759
Title: A Phase 2, Multicenter, Double- Blind, Parallel-group, Randomized, Placebo-controlled, Forced-dose Titration, Dose-ranging Efficacy and Safety Study of SPD489 in Combination With an Antidepressant in the Treatment of Adults With Major Depressive Disorder With Inadequate Response to Prospective Treatment With an Antidepressant
Brief Title: SPD489 in Combination With an Antidepressant in the Treatment of Adults With Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPD489-209; 2011-003615-28 (EudraCT Number)
Record Dates: First submitted 2011-09-15; First posted 2011-09-19 (Estimated); Results first posted 2015-02-19 (Estimated); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Antidepressive Agents; Lisdexamfetamine Dimesylate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (5):
- Antidepressant + SPD489 10 mg (Experimental)
  Interventions: Drug: Antidepressant + SPD489 (Lisdexamfetamine dimesylate) 10 mg
- Antidepressant + SPD489 30 mg (Experimental)
  Interventions: Drug: Antidepressant + SPD489 (Lisdexamfetamine dimesylate) 30 mg
- Antidepressant + SPD489 50 mg (Experimental)
  Interventions: Drug: Antidepressant + SPD489 (Lisdexamfetamine dimesylate) 50 mg
- Antidepressant + SPD489 70 mg (Experimental)
  Interventions: Drug: Antidepressant + SPD489 (Lisdexamfetamine dimesylate) 70 mg
- Antidepressant + Placebo (Placebo Comparator)
  Interventions: Drug: Antidepressant + Placebo

INTERVENTIONS:
Drug: Antidepressant + SPD489 (Lisdexamfetamine dimesylate) 10 mg — Antidepressant + SPD489 oral, 10 mg, once daily for 8 weeks
  Other Names: Vyvanse
  Arms: Antidepressant + SPD489 10 mg
Drug: Antidepressant + SPD489 (Lisdexamfetamine dimesylate) 30 mg — Antidepressant + SPD489 oral, 30 mg, once daily for 8 weeks
  Other Names: Vyvanse
  Arms: Antidepressant + SPD489 30 mg
Drug: Antidepressant + SPD489 (Lisdexamfetamine dimesylate) 50 mg — Antidepressant + SPD489 oral, 50 mg, once daily for 8 weeks
  Other Names: Vyvanse
  Arms: Antidepressant + SPD489 50 mg
Drug: Antidepressant + SPD489 (Lisdexamfetamine dimesylate) 70 mg — Antidepressant + SPD489 oral, 70 mg, once daily for 8 weeks
  Other Names: Vyvanse
  Arms: Antidepressant + SPD489 70 mg
Drug: Antidepressant + Placebo — oral, once daily for 8 weeks
  Arms: Antidepressant + Placebo

SUMMARY:
This study will examine SPD489 in subjects aged 18-65 with major depressive disorder (MDD) who are taking certain types of antidepressants but continue to have residual depression symptoms. The purpose of this study is to help answer the following questions:

* How safe is SPD489 for the supplemental treatment of depression and what are the side effects that might be related to it?
* Can SPD489 help patients with depression who are also taking an antidepressant?
* How much SPD489 should be given to patients with depression who are also taking an antidepressant?
* How does SPD489 compare to placebo in depressed patients who are also taking an antidepressant?

ELIGIBILITY:
Inclusion Criteria

1. Subject is able to provide written, personally signed and dated informed consent to participate in the study before completing any study-related procedures.
2. Subject is between 18-65 years of age.
3. Subject has a primary diagnosis of non-psychotic MDD.
4. Subject has a MADRS total score 24
5. Subject is willing and has an understanding and ability to fully comply with study procedures and restrictions defined in this protocol.
6. Subject, who is female, must have a negative serum beta human chorionic gonadotropin (HCG) pregnancy test and a negative urine pregnancy test and agrees to comply with any applicable contraceptive requirements.
7. Subject is able to swallow a capsule.

Exclusion Criteria

1. Subject whose current episode of MDD has not responded to an adequate treatment regimen.
2. Subject who has a lifetime history of treatment resistant depression, defined as having not responded to adequate treatment with 2 or more treatment regimens.
3. Subject has a current comorbid psychiatric disorder that is either controlled with medications prohibited in this study or is uncontrolled and associated with significant symptoms.
4. Subject has been hospitalized (within the last 12 months) for their current MDD episode.
5. Subject has a current or lifetime history of attention-deficit/hyperactivity disorder (ADHD).
6. Subject has a first degree relative that has been diagnosed with bipolar I disorder.
7. Subject has a recent history (within the last 6 months) of suspected substance abuse or dependence disorder.
8. Subject is considered a suicide risk, has previously made a suicide attempt within the past 3 years, or is currently demonstrating active suicidal ideation.
9. Subject has a concurrent chronic or acute illness or unstable medical condition.
10. Subject has a history of seizures (other than infantile febrile seizures), any tic disorder, or a current diagnosis and/or a known family history of Tourette's Disorder, serious neurological disease, history of significant head trauma, dementia, cerebrovascular disease, Parkinson's disease, or intracranial lesions.
11. Subject has known history of symptomatic cardiovascular disease, advanced arteriosclerosis, structural cardiac abnormality, cardiomyopathy, serious heart rhythm abnormalities, coronary artery disease, or other serious cardiac problems that may place them at increased vulnerability to the sympathomimetic effects of a stimulant medication.
12. Subject has a history of thyroid disorder that has not been stabilized on thyroid medication or treatment within 3 months prior to the Screening Visit.
13. Subject has a known family history of sudden cardiac death or ventricular arrhythmia.
14. Subject has glaucoma.
15. Subject has any clinically significant ECG or clinical laboratory abnormalities at the Screening Visit.
16. Subject has a history of moderate to severe hypertension.
17. Current use of any other medication (including over-the-counter [OTC], herbal or homeopathic preparations) that has central nervous system effects.
18. Subject has the potential to need to initiate or modify frequency of psychotherapy or to continue or initiate other treatments for depression, outside of those allowed in this protocol.
19. Subject has had electroconvulsive therapy for the current depressive episode 3 months prior to the Lead-in Baseline Visit.
20. The subject has a known or suspected intolerance or hypersensitivity to the investigational product.
21. The subject has a known or suspected intolerance or hypersensitivity to any of the possible antidepressant treatments (escitalopram oxalate or venlafaxine HCL extended release.
22. Subject has a positive urine drug result.
23. Subject has a body mass index of <18.5 or >40.
24. Subject is female and is pregnant or nursing.
25. Subject has participated in another clinical study involving SPD489/NRP104 or has previously used commercial lisdexamfetamine dimesylate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1197 (Actual)
Dates: Start 2011-05-31 (Actual); Primary Completion 2014-01-17 (Actual); Study Completion 2014-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (82):
- United States (60):
  - Arkansas Psychiatric Clinic Clinical Research Trials, Little Rock, Arkansas
  - South Coast Clinical Trials, Anaheim, California
  - Catalina Research Institute, LLC, Chino, California
  - Shanti Clinical Trials, Colton, California
  - Clinical Innovation, Inc., Costa Mesa, California
  - Collaborative Neuroscience Network, Inc., Garden Grove, California
  - Irvine Center for Clinical Research, Irvine, California
  - Omega Clinical Trials, La Habra, California
  - Provate Practice of Andrew Leuchter, MD, Los Angeles, California
  - PCSD - Feighner Research, San Diego, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Neuropsychiatric Research Center of Orange County, Santa Ana, California
  - California Neuroscience Research Medical Group, Inc., Sherman Oaks, California
  - Western Affiliated Research Institute, Denver, Colorado
  - Connecticut Clinical Research, Cromwell, Connecticut
  - Institute of Living, Hartford, Connecticut
  - The Hospital of Central Connecticut, Psychiatry & Behavioral Health Research, New Britain, Connecticut
  - Gulfcoast Clinical Research Center, Fort Myers, Florida
  - Sarkis Clinical Trials, Gainesville, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Private Practice - Amit Vijapura MD, Jacksonville, Florida
  - Psychiatric Associates, Lake City, Florida
  - Comprehensive Neuroscience, Inc., Miramar, Florida
  - Fideltiy Clinical Research, Inc., North Miami, Florida
  - Ali A. Kashfi, MD, PA, Orlando, Florida
  - Clinical Research of Central Florida, Winter Haven, Florida
  - Kolin Research Group, Winter Park, Florida
  - Institute for Behavioral Medicine, LLC, Smyrna, Georgia
  - Treatment Research Center, Rush University Medical Center, Chicago, Illinois
  - Alexian Brothers Center for Psychiatric Research, Hoffman Estates, Illinois
  - Psychiatric Medicine Associates, LLC, Skokie, Illinois
  - Sleep and Behavior Medicine Institute, Vernon Hills, Illinois
  - Clinical Trials Technology, Inc., Prairie Village, Kansas
  - Pedia Research, LLC, Owensboro, Kentucky
  - Psyichatric Care and Research Center, O'Fallon, Missouri
  - Mid-America Clinical Research, LLC, St Louis, Missouri
  - Premier Psychiatric Research Institute, LLC., Lincoln, Nebraska
  - Clinical Research Consortium, Las Vegas, Nevada
  - Center for Emotional Fitness, Cherry Hill, New Jersey
  - CRI Worldwide LLC, Willingboro, New Jersey
  - Albuquerque Neuroscience, Inc., Albuquerque, New Mexico
  - Clinlabs, Inc., New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Private Practice - Daniel I. Rifkin MD PC, West Seneca, New York
  - Clinical Trials of America, Inc., Hickory, North Carolina
  - North Coast Clinical Trials, Inc., Beachwood, Ohio
  - Ohio State University, Dept. of Psychiatry, Columbus, Ohio
  - Neurology & Neuroscience Center of Ohio, Toledo, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University Services, West Chester, Pennsylvania
  - Pillar Clinical Research, LLC, Dallas, Texas
  - Bay Area Clinical Services, Friendswood, Texas
  - Houston Clinical Trials, LLC, Houston, Texas
  - Wharton Research Center, Inc., Wharton, Texas
  - Grayline Clinical Drug Trials, Wichita Falls, Texas
  - Alliance Research Group, Richmond, Virginia
  - Dean Foundation for Health, Research and Education, Inc., Middleton, Wisconsin
  - Independent Psychiatric Consultants, SC, dba, IPC Research, Waukesha, Wisconsin
- Argentina (5):
  - Instituto Nacional de Psicopatologia, Buenos Aires
  - Cervino, Buenos Aires
  - Centro Medico de Medicina Familiar Mind Out Research, CABA
  - BA Psychiatric Research Center, CABA
  - Instituto Medico SAMIC, Córdoba
- Australia (5):
  - Peninsula Health Mental Health Services, Frankston, Victoria
  - Neurotherapy Victoria, Malvern, Victoria
  - The Alfred, Monash Alfred Psychiatry Research Centre, Melbourne, Victoria
  - The Melbourne Clinic, Richmond, Victoria
  - Lyell McEwin Hospital, Mental Health Clinical Trials Unit, Elizabeth Vale
- Chile (7):
  - Psocomed Estudios Medicos, Antofagasta, Il Region
  - Especialidades Medicas L y S, Las Condes, Santiago Metropolitan
  - Centro de Estudios y Tratemiento de Enfermedades Psiquiatricas, Las Condes, Santiago Metropolitan
  - Biomedica Research Group, Providencia, Santiago Metropolitan
  - Centro de Estudios Clinicos, Providencia, Santiago Metropolitan
  - Unidad de Salud Mental y Psiquietriea Hospital y CRS El Pino, San Bernardo, Santiago Metropolitan
  - Hospital Barros Luco Trudsau, San Miguel, Santiago Metropolitan
- United Kingdom (5):
  - Hollins Park Hospital, Winwick, Warrington Cheshire
  - Radbourne Unit, Derby
  - ADHD Mental Health Research Unit, Horsham
  - Newcastle University, Wolfson Research Centre, Newcastle upon Tyne
  - Rushcliffe Mental Health Team, Nottingham

REFERENCES:
- [Result] Richards C, Iosifescu DV, Mago R, Sarkis E, Reynolds J, Geibel B, Dauphin M. A randomized, double-blind, placebo-controlled, dose-ranging study of lisdexamfetamine dimesylate augmentation for major depressive disorder in adults with inadequate response to antidepressant therapy. J Psychopharmacol. 2017 Sep;31(9):1190-1203. doi: 10.1177/0269881117722998. Epub 2017 Aug 31. PMID 28857719

RESULTS

PARTICIPANT FLOW:
Groups:
- Antidepressant + Single-blind Placebo: Subjects received unblinded standard antidepressant therapy (either escitalopram oxalate or venlafaxine hydrochloride extended-release titrated to the maximum tolerated dose) plus oral, once daily single-blind placebo (matching SPD489).
- Antidepressant + Double-blind Placebo: Subjects received unblinded standard antidepressant therapy (either escitalopram oxalate or venlafaxine hydrochloride extended-release titrated to the maximum tolerated dose) plus oral, once daily double-blind placebo (matching SPD489).
- Antidepressant + Double-blind SPD489 10mg: Subjects received unblinded standard antidepressant therapy (either escitalopram oxalate or venlafaxine hydrochloride extended-release titrated to the maximum tolerated dose) plus oral, once daily over-encapsulated SPD489 as a 10mg dose.
- Antidepressant + Double-blind SPD489 30mg: Subjects received unblinded standard antidepressant therapy (either escitalopram oxalate or venlafaxine hydrochloride extended-release titrated to the maximum tolerated dose) plus oral, once daily over-encapsulated SPD489 as a 30mg dose.
- Antidepressant + Double-blind SPD489 50mg: Subjects received unblinded standard antidepressant therapy (either escitalopram oxalate or venlafaxine hydrochloride extended-release titrated to the maximum tolerated dose) plus oral, once daily over-encapsulated SPD489 as a 50mg dose.
- Antidepressant + Double-blind SPD489 70mg: Subjects received unblinded standard antidepressant therapy (either escitalopram oxalate or venlafaxine hydrochloride extended-release titrated to the maximum tolerated dose) plus oral, once daily over-encapsulated SPD489 as a 70mg dose.
Period: Antidepressant Lead-in Phase
Arm/Group | Antidepressant + Single-blind Placebo | Antidepressant + Double-blind Placebo | Antidepressant + Double-blind SPD489 10mg | Antidepressant + Double-blind SPD489 30mg | Antidepressant + Double-blind SPD489 50mg | Antidepressant + Double-blind SPD489 70mg
Started | 1197 (Of these 1197 subjects, 19 subjects were not dosed.) | 0 | 0 | 0 | 0 | 0
Completed | 855 | 0 | 0 | 0 | 0 | 0
Not Completed | 342 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 40 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 16 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 74 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 83 | 0 | 0 | 0 | 0 | 0
Not completed — Met BP or Pulse Withdrawal Criteria | 10 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 119 | 0 | 0 | 0 | 0 | 0
Period: Double-blind Phase
Arm/Group | Antidepressant + Single-blind Placebo | Antidepressant + Double-blind Placebo | Antidepressant + Double-blind SPD489 10mg | Antidepressant + Double-blind SPD489 30mg | Antidepressant + Double-blind SPD489 50mg | Antidepressant + Double-blind SPD489 70mg
Started | 463 (These subjects were not included in the Safety Dose Response Evaluable Set or Safety Analysis Set.) | 78 | 78 (One subject was not dosed.) | 78 (Two subjects were not dosed.) | 78 | 80
Completed | 397 | 71 | 71 | 69 | 69 | 71
Not Completed | 66 | 7 | 7 | 9 | 9 | 9
Not completed — Adverse Event | 7 | 0 | 1 | 1 | 1 | 3
Not completed — Protocol Violation | 2 | 0 | 1 | 2 | 0 | 1
Not completed — Withdrawal by Subject | 17 | 4 | 3 | 4 | 2 | 2
Not completed — Lost to Follow-up | 31 | 1 | 2 | 0 | 3 | 3
Not completed — Met BP or Pulse Withdrawal Criteria | 1 | 0 | 0 | 0 | 3 | 0
Not completed — Other | 8 | 2 | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: All subjects who took at least 1 dose of randomized investigational product and who had at least 1 post-augmentation baseline safety assessment (e.g. coming back for any visit, reporting of an adverse event [AE] or reporting the absence of AEs). Subjects who received only single-blind placebo were not included in this group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Antidepressant + Double-blind Placebo | Antidepressant + Double-blind SPD489 10mg | Antidepressant + Double-blind SPD489 30mg | Antidepressant + Double-blind SPD489 50mg | Antidepressant + Double-blind SPD489 70mg | Total
Number analyzed (Participants) | 78 | 77 | 76 | 78 | 80 | 389
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.7 (10.48) | 39.1 (11.83) | 43.4 (12.06) | 43.8 (12.4) | 41.5 (10.81) | 42.3 (11.61)
Age, Customized [Count of Participants; unit: Participants]
  18-55 | 69 | 70 | 62 | 60 | 71 | 332
  56-65 | 9 | 7 | 14 | 18 | 9 | 57
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 53 | 52 | 53 | 53 | 264
  Male | 25 | 24 | 24 | 25 | 27 | 125
Region of Enrollment [Count of Participants; unit: Participants]
  ARGENTINA | 2 | 3 | 5 | 3 | 5 | 18
  AUSTRALIA | 0 | 0 | 0 | 2 | 3 | 5
  CHILE | 3 | 6 | 12 | 9 | 2 | 32
  UNITED KINGDOM | 1 | 0 | 0 | 0 | 0 | 1
  UNITED STATES | 72 | 68 | 59 | 64 | 70 | 333

OUTCOME MEASURES:

1. Secondary Outcome: Change in Average Systolic Blood Pressure From Augmentation Baseline (Week 8) to Week 16
Time Frame: From Augmentation Baseline (Week 8) to Week 16
Population: Vital Signs Evaluable Set: All randomized subjects who had at least 1 valid vital signs measurement during the Dose Maintenance Period while on the target dose level of investigational product.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Antidepressant + Double-blind Placebo | Antidepressant + Double-blind SPD489 10mg | Antidepressant + Double-blind SPD489 30mg | Antidepressant + Double-blind SPD489 50mg | Antidepressant + Double-blind SPD489 70mg
Number analyzed (Participants) | 67 | 68 | 65 | 51 | 63
mmHg | -0.2 (9.55) | 0.2 (8.58) | 0.5 (9.17) | 3.5 (7.82) | 2.6 (10.55)
Statistical Analysis 1: Comparison: Antidepressant + Double-blind Placebo vs Antidepressant + Double-blind SPD489 10mg vs Antidepressant + Double-blind SPD489 30mg vs Antidepressant + Double-blind SPD489 50mg vs Antidepressant + Double-blind SPD489 70mg; Test type: Superiority or Other; p = 0.004, MCP-Mod Analysis; The systolic blood pressure p-value was based on a critical value of 1.99 from a multivariate-t distribution with 341 degrees of freedom; Least Squares Mean = 3.16, Standard Error of Mean 1.01 — The t-statistic used for this analysis, 3.14, was based on MCP-Mod Analysis for the candidate model EMax
Statistical Analysis 2: Comparison: Antidepressant + Double-blind Placebo vs Antidepressant + Double-blind SPD489 10mg vs Antidepressant + Double-blind SPD489 30mg vs Antidepressant + Double-blind SPD489 50mg vs Antidepressant + Double-blind SPD489 70mg; Test type: Superiority or Other; p = 0.032, MCP-Mod Analysis; [statistical method as in outcome 1, analysis 1]; Least Squares Means = 2.50, Standard Error of Mean 1.01 — The t-statistic used for this analysis, 2.48, was based on MCP-Mod Analysis for the candidate model Exponential
Statistical Analysis 3: Comparison: Antidepressant + Double-blind Placebo vs Antidepressant + Double-blind SPD489 10mg vs Antidepressant + Double-blind SPD489 30mg vs Antidepressant + Double-blind SPD489 50mg vs Antidepressant + Double-blind SPD489 70mg; Test type: Superiority or Other; p = 0.003, MCP-Mod Analysis; [statistical method as in outcome 1, analysis 1]; Least Squares Mean = 3.28, Standard Error of Mean 1.01 — The t-statistic used for this analysis, 3.26 was based on MCP-Mod Analysis for the candidate model Linear
Statistical Analysis 4: Comparison: Antidepressant + Double-blind Placebo vs Antidepressant + Double-blind SPD489 10mg vs Antidepressant + Double-blind SPD489 30mg vs Antidepressant + Double-blind SPD489 50mg vs Antidepressant + Double-blind SPD489 70mg; Test type: Superiority or Other; p = 0.010, MCP-Mod Analysis Method; [statistical method as in outcome 1, analysis 1]; Least Squares Means = 2.91, Standard Error of Mean 1.01 — The t-statistic used for this analysis, 2.88, was based on MCP-Mod Analysis for the candidate model Logistic1
Statistical Analysis 5: Comparison: Antidepressant + Double-blind Placebo vs Antidepressant + Double-blind SPD489 10mg vs Antidepressant + Double-blind SPD489 30mg vs Antidepressant + Double-blind SPD489 50mg vs Antidepressant + Double-blind SPD489 70mg; Test type: Superiority or Other; p = 0.005, MCP-Mod Analysis; [statistical method as in outcome 1, analysis 1]; Least Squares Means = 3.15, Standard Error of Mean 1.01 — The t-statistic used for this analysis, 3.12, was based on MCP-Mod Analysis for the candidate model Logistic2

2. Secondary Outcome: Change in Average Diastolic Blood Pressure From Augmentation Baseline (Week 8) to Week 16
Time Frame: From Augmentation Baseline (Week 8) to Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Antidepressant + Double-blind Placebo | Antidepressant + Double-blind SPD489 10mg | Antidepressant + Double-blind SPD489 30mg | Antidepressant + Double-blind SPD489 50mg | Antidepressant + Double-blind SPD489 70mg
Number analyzed (Participants) | 67 | 68 | 65 | 51 | 63
mmHg | -0.1 (6.69) | -0.9 (6.64) | -0.1 (7.39) | 2.8 (6.58) | 1.9 (7.45)
Statistical Analysis 1: Comparison: Antidepressant + Double-blind Placebo vs Antidepressant + Double-blind SPD489 10mg vs Antidepressant + Double-blind SPD489 30mg; Test type: Superiority or Other; p = 0.011, MCP-Mod Analysis; The diastolic blood pressure p-value was based on a critical value of 1.99 from a multivariate-t distribution with 341 degrees of freedom; Least Squares Means = 2.16, Standard Error of Mean 0.75 — The t-statistic used for this analysis, 2.86 was based on MCP-Mod Analysis for the candidate model Emax
Statistical Analysis 2: Comparison: Antidepressant + Double-blind Placebo vs Antidepressant + Double-blind SPD489 10mg vs Antidepressant + Double-blind SPD489 30mg vs Antidepressant + Double-blind SPD489 50mg vs Antidepressant + Double-blind SPD489 70mg; Test type: Superiority or Other; p = 0.023, MCP-Mod Analysis; [statistical method as in outcome 2, analysis 1]; Least Squares Means = 1.95, Standard Error of Mean 0.75 — The t-statistic used for this analysis, 2.59, was based on MCP-Mod Analysis for the candidate model Exponential
Statistical Analysis 3: Comparison: Antidepressant + Double-blind Placebo vs Antidepressant + Double-blind SPD489 10mg vs Antidepressant + Double-blind SPD489 30mg vs Antidepressant + Double-blind SPD489 50mg vs Antidepressant + Double-blind SPD489 70mg; Test type: Superiority or Other; p = 0.003, Least Squares Means; [statistical method as in outcome 2, analysis 1]; MCP-Mod Analysis = 2.47, Standard Error of Mean 0.75 — The t-statistic used for this analysis, 3.28, was based on MCP-Mod Analysis for the candidate model Linear
Statistical Analysis 4: Comparison: Antidepressant + Double-blind Placebo vs Antidepressant + Double-blind SPD489 10mg vs Antidepressant + Double-blind SPD489 30mg vs Antidepressant + Double-blind SPD489 50mg vs Antidepressant + Double-blind SPD489 70mg; Test type: Superiority or Other; p = 0.009, MCP-Mod Analysis; [statistical method as in outcome 2, analysis 1]; Least Squares Means = 2.22, Standard Error of Mean 0.76 — The t-statistic used for this analysis, 2.93, was based on MCP-Mod Analysis for the candidate model Logistic1
Statistical Analysis 5: Comparison: Antidepressant + Double-blind Placebo vs Antidepressant + Double-blind SPD489 10mg vs Antidepressant + Double-blind SPD489 30mg vs Antidepressant + Double-blind SPD489 50mg vs Antidepressant + Double-blind SPD489 70mg; Test type: Superiority or Other; p = 0.005, MCP-Mod Analysis; [statistical method as in outcome 2, analysis 1]; Least Squares Means = 2.37, Standard Error of Mean 0.76 — The t-statistic used for this analysis, 3.13, was based on MCP-Mod Analysis for the candidate model Logistic2

3. Secondary Outcome: Change in Average Pulse Rate From Augmentation Baseline (Week 8) to Week 16
Time Frame: From Augmentation Baseline (Week 8) to Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Antidepressant + Double-blind Placebo | Antidepressant + Double-blind SPD489 10mg | Antidepressant + Double-blind SPD489 30mg | Antidepressant + Double-blind SPD489 50mg | Antidepressant + Double-blind SPD489 70mg
Number analyzed (Participants) | 67 | 68 | 65 | 51 | 63
bpm | -0.8 (9.95) | 0.8 (7.32) | 5.3 (8.08) | 4.0 (9.80) | 6.0 (11.25)
Statistical Analysis 1: Comparison: Antidepressant + Double-blind Placebo vs Antidepressant + Double-blind SPD489 10mg vs Antidepressant + Double-blind SPD489 30mg vs Antidepressant + Double-blind SPD489 50mg vs Antidepressant + Double-blind SPD489 70mg; Test type: Superiority or Other; p < 0.001, MCP-Mod Analysis; The pulse p-value was based on a critical value of 1.99 from a multivariate-t distribution with 341 degrees of freedom; Least Squares Means = 4.45, Standard Error of Mean 1.05 — The t-statistic used for this analysis, 4.24, was based on MCP-Mod Analysis for the candidate model Emax
Statistical Analysis 2: Comparison: Antidepressant + Double-blind Placebo vs Antidepressant + Double-blind SPD489 10mg vs Antidepressant + Double-blind SPD489 30mg vs Antidepressant + Double-blind SPD489 50mg vs Antidepressant + Double-blind SPD489 70mg; Test type: Superiority or Other; p = 0.002, MCP-Mod Analysis; The pulse p-value was based on a critical value of 1.99 from a multivariate-t distribution with 341 degrees of freedom; Least Squares Means = 3.52, Standard Error of Mean 1.05 — The t-statistic used for this analysis, 3.36, was based on MCP-Mod Analysis for the candidate model Expontential
Statistical Analysis 3: Comparison: Antidepressant + Double-blind Placebo vs Antidepressant + Double-blind SPD489 10mg vs Antidepressant + Double-blind SPD489 30mg vs Antidepressant + Double-blind SPD489 50mg vs Antidepressant + Double-blind SPD489 70mg; Test type: Superiority or Other; p < 0.001, MCP-Mod Analysis; The pulse p-value was based on a critical value of 1.99 from a multivariate-t distribution with 341 degrees of freedom; Least Squares Means = 4.30, Standard Error of Mean 1.05 — The t-statistic used for this analysis, 4.10, was based on MCP-Mod Analysis for the candidate model Linear
Statistical Analysis 4: Comparison: Antidepressant + Double-blind Placebo vs Antidepressant + Double-blind SPD489 10mg vs Antidepressant + Double-blind SPD489 30mg vs Antidepressant + Double-blind SPD489 50mg vs Antidepressant + Double-blind SPD489 70mg; Test type: Superiority or Other; p < 0.001, MCP-Mod Analysis; The pulse p-value was based on a critical value of 1.99 from a multivariate-t distribution with 341 degrees of freedom; Least Squares Means = 4.63, Standard Error of Mean 1.05 — The t-statistic used for this analysis, 4.39, was based on MCP-Mod Analysis for the candidate model Logistic1
Statistical Analysis 5: Comparison: Antidepressant + Double-blind Placebo vs Antidepressant + Double-blind SPD489 10mg vs Antidepressant + Double-blind SPD489 30mg vs Antidepressant + Double-blind SPD489 50mg vs Antidepressant + Double-blind SPD489 70mg; Test type: Superiority or Other; p < 0.001, MCP-Mod Analysis; The pulse p-value was based on a critical value of 1.99 from a multivariate-t distribution with 341 degrees of freedom; Least Squares Means = 4.63, Standard Error of Mean 1.05 — The t-statistic used for this analysis, 4.39 was based on MCP-Mod Analysis for the candidate model Logistic2

4. Primary Outcome: Change in Montgomery-Ǻsberg Depression Rating Scale (MADRS) Total Score From Augmentation Baseline (Week 8) to Week 16 (Double-blind Phase, Dose Response Evaluable Set)
Description: MADRS is a validated, 10-item rating scale with each item being scored on a scale from 0-6 with a total score ranging from 0-60. Lower scores indicate a decreased severity of depression. CHange in MADRS total score in Augmentsion Baseline to Week 16.
Time Frame: Augmentation Baseline (Week 8) to Week 16
Population: Dose Response Evaluable Set (DRES): All randomized subjects who had at least 1 valid primary efficacy measurement (MADRS total score) during the Dose Maintenance Period (Weeks 11-16) while on the target dose level of investigational product.
Measure: Least Squares Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | Antidepressant + Double-blind Placebo | Antidepressant + Double-blind SPD489 10mg | Antidepressant + Double-blind SPD489 30mg | Antidepressant + Double-blind SPD489 50mg | Antidepressant + Double-blind SPD489 70mg
Number analyzed (Participants) | 72 | 71 | 69 | 66 | 71
units on a scale | -5.4 [-7.2 to -3.5] | -6.7 [-8.6 to -4.9] | -5.3 [-7.1 to -3.4] | -6.1 [-8.1 to -4.1] | -6.3 [-8.2 to -4.4]
Statistical Analysis 1: Comparison: Antidepressant + Double-blind Placebo vs Antidepressant + Double-blind SPD489 10mg vs Antidepressant + Double-blind SPD489 30mg vs Antidepressant + Double-blind SPD489 50mg vs Antidepressant + Double-blind SPD489 70mg; Analysis of Dose-Response Using the MCP-Mod Analysis Method; Test type: Superiority or Other; p = 1.000, MCP-Mod Analysis Method — Any p-value <=0.10 indicates successful establishment of dose-response relationship; The adjusted p-value was based on a critical value of 2.02 from a multivariate-t distribution with 341 degrees of freedom; Least Squares Means = -.11, Standard Error of Mean 1.07 — The t-statistic used for this analysis, 0.10, was based on MCP-Mod Analysis from the linear contrast using optimal coefficients for the pre-specified candidate model Betamod
Statistical Analysis 2: Comparison: Antidepressant + Double-blind Placebo vs Antidepressant + Double-blind SPD489 10mg vs Antidepressant + Double-blind SPD489 30mg vs Antidepressant + Double-blind SPD489 50mg vs Antidepressant + Double-blind SPD489 70mg; Analysis of Dose-Response Using the MCP-Mod Analysis Method; Test type: Superiority or Other; p = 0.942, MCP-Mod Analysis — Any p-value <=0.10 indicates successful establishment of dose-response relationship; [statistical method as in outcome 4, analysis 1]; Least Squares Means = 0.43, Standard Error of Mean 1.06 — The t-statistic used for this analysis, 0.41, was based on MCP-Mod Analysis from the linear contrast using optimal coefficients for the pre-specified candidate model Emax
Statistical Analysis 3: Comparison: Antidepressant + Double-blind Placebo vs Antidepressant + Double-blind SPD489 10mg vs Antidepressant + Double-blind SPD489 30mg vs Antidepressant + Double-blind SPD489 50mg vs Antidepressant + Double-blind SPD489 70mg; Analysis of Dose-Response Using the MCP-Mod Analysis Method; Test type: Superiority or Other; p = 0.995, MCP-Mod Analysis — Any p-value <=0.10 indicates successful establishment of dose-response relationship; [statistical method as in outcome 4, analysis 1]; Least Squares Means = 0.21, Standard Error of Mean 1.06 — The t-statistic used for this analysis, 0.20, was based on MCP-Mod Analysis from the linear contrast using optimal coefficients for the pre-specified candidate model Linear
Statistical Analysis 4: Comparison: Antidepressant + Double-blind Placebo vs Antidepressant + Double-blind SPD489 10mg vs Antidepressant + Double-blind SPD489 30mg vs Antidepressant + Double-blind SPD489 50mg vs Antidepressant + Double-blind SPD489 70mg; Analysis of Dose-Response Using the MCP-Mod Analysis Method; Test type: Superiority or Other; p = 0.978, MCP-Mod Analysis — Any p-value <=0.10 indicates successful establishment of dose-response relationship; [statistical method as in outcome 4, analysis 1]; Least Squares Means = -.32, Standard Error of Mean 1.07 — The t-statistic used for this analysis, 0.30, was based on MCP-Mod Analysis from the linear contrast using optimal coefficients for the pre-specified candidate model Logistic

ADVERSE EVENTS:
Description: Safety Analysis Set: All subjects who took at least 1 dose of randomized investigational product and who had at least 1 post-augmentation baseline safety assessment (e.g. coming back for any visit, reporting of an AE or reporting the absence of AEs). Subjects who received only single-blind placebo were not included in this group.
Arm/Group | Antidepressant + Double-blind Placebo | Antidepressant + Double-blind SPD489 10mg | Antidepressant + Double-blind SPD489 30mg | Antidepressant + Double-blind SPD489 50mg | Antidepressant + Double-blind SPD489 70mg
Serious Adverse Events (participants affected / at risk) | 0/78 | 0/77 | 0/76 | 0/78 | 1/80
Other Adverse Events (participants affected / at risk) | 20/78 | 30/77 | 29/76 | 36/78 | 44/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Antidepressant + Double-blind Placebo (N=78) | Antidepressant + Double-blind SPD489 10mg (N=77) | Antidepressant + Double-blind SPD489 30mg (N=76) | Antidepressant + Double-blind SPD489 50mg (N=78) | Antidepressant + Double-blind SPD489 70mg (N=80)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Antidepressant + Double-blind Placebo (N=78) | Antidepressant + Double-blind SPD489 10mg (N=77) | Antidepressant + Double-blind SPD489 30mg (N=76) | Antidepressant + Double-blind SPD489 50mg (N=78) | Antidepressant + Double-blind SPD489 70mg (N=80)
Diarrhoea (Gastrointestinal disorders) | 4 (5) | 2 (2) | 3 (3) | 2 (2) | 5 (5)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 10 (10) | 10 (10)
Nausea (Gastrointestinal disorders) | 1 (1) | 5 (5) | 6 (6) | 1 (1) | 6 (7)
Fatigue (General disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 4 (4)
Influenza (Infections and infestations) | 2 (3) | 1 (1) | 4 (4) | 4 (5) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 5 (5) | 4 (5) | 2 (2) | 7 (8)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3) | 3 (3) | 4 (4) | 3 (3)
Urinary tract infection (Infections and infestations) | 5 (5) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 4 (4) | 5 (6) | 5 (5) | 4 (6)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2) | 2 (2) | 5 (5) | 1 (1)
Headache (Nervous system disorders) | 10 (12) | 7 (8) | 5 (9) | 3 (5) | 8 (9)
Bruxism (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 6 (7)
Insomnia (Psychiatric disorders) | 2 (2) | 7 (9) | 2 (2) | 8 (10) | 9 (11)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.